CLINICAL TRIAL: NCT01287104
Title: A Phase I Study of NK Cell Infusion Following Allogeneic Peripheral Blood Stem Cell Transplantation From Related or Matched Unrelated Donors in Pediatric Patients With Hematologic Malignancies
Brief Title: A Phase I Study of NK Cell Infusion Following Allogeneic Peripheral Blood Stem Cell Transplantation From Related or Matched Unrelated Donors in Pediatric Patients With Solid Tumors and Leukemias
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Nirali N. Shah, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 110073; 11-C-0073
Record Dates: First submitted 2011-01-29; First posted 2011-02-01 (Estimated); Results first posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Leukemia; Lymphoma
Keywords: Leukemia/Lymphoma; Hematologic Malignancies; Leukemia; Lymphoma; Ewing Sarcoma; Rhabdomyosarcoma; Neuroblastoma; Healthy Donor
MeSH Terms: conditions — Leukemia; Lymphoma; Hematologic Neoplasms; Sarcoma, Ewing; Rhabdomyosarcoma; Neuroblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pre-Bone Marrow Transplant (BMT) Prep Regimen (Experimental): Pre-bone marrow transplant (BMT) Prep Regimen with Stem Cell and natural killer (NK) Cell Infusions coupled with Induction therapy
  Interventions: Biological: Natural Killer (NK) Cell Infusion; Biological: Stem Cell Infusion

INTERVENTIONS:
Biological: Natural Killer (NK) Cell Infusion — Post-transplant Day 21 (plus-minus 3 days): (1 x 10(5), 1 x 10(6) or 1 x 10(7) natural killer (NK) cells/kg by intravenous (IV) infusion. Followed by a second NK cell infusion of the same cell dose, on Day 49 plus-minus 7 days.
Biological: Stem Cell Infusion — Transplant Day 0: >4 x 10(6)/kg cluster of differentiation 34 (CD34)+ stem cells by IV infusion Filgrastim, 5 microgram/kg per day subcutaneous (SQ) from day 0 until absolute neutrophil count (ANC) >5000/microliters x2

SUMMARY:
Background:

* Bone marrow stem cells, which are found in the bone marrow and blood stream, can be collected and transplanted to treat a variety of types of cancer in a process known as hematopoietic stem cell transplantation (HSCT). When stem cells are taken from one person, most commonly a sibling or a family member, and then given to another person, this is referred to as allogeneic HSCT. Allogeneic HSCT has proven to be an especially effective treatment for patients with some types of cancers of the blood (leukemia) and certain solid tumors. The transplanted stem cells travel to the patient's bone marrow and begin producing normal blood cells, and also attack patients cancer cells.
* Because allogenic HSCT does not always prevent the cancer from returning, researchers are interested in determining whether another type of immune cell taken from the stem cell donors white blood cells, called a "natural killer" (NK) cell, can be given in addition to the HSCT to help fight the tumor. In the laboratory, NK cells have been shown to kill tumor cells, but it is not yet know if this will occur when given to patients after HSCT.

Objectives:

* To determine the safety, effectiveness, and immune system response of giving NK white blood cells to individuals who have received allogeneic HSCT.
* To identify possible side effects from the treatment.

Eligibility:

* Donors: Stem cell donors whose blood matches one of the recipients on six out of six human leukocyte antigen (HLA) (blood immune marker) types. The donor may not be the identical twin of a recipient.
* Recipients: Individuals between 4 and 35 years of age who have been diagnosed with pediatric solid tumors that have not responded to standard treatment, or individuals between 4 and 18 years of age who have been diagnosed with leukemia that has not responded to standard treatment.
* Other eligibility requirements which include a physical exam and blood laboratory evaluation are included to make sure it is safe for both the donor to donate and the recipient to undergo the transplant procedure.

Design:

* Donors and recipients will be screened with a full medical history and physical examination, and will provide blood and urine samples; recipients will have tumor imaging studies and other tests as required by the researchers.
* Donors:
* Participants will receive filgrastim injections (to stimulate the bone marrow) for 1 week to make stem cells travel from bone marrow to blood.
* Participants will provide stem cells and NK cells through apheresis.
* Recipients:
* Participants will have three cycles of chemotherapy to treat the underlying cancer and weaken the immune system so that it will accept the donor cells.
* Participants will then receive preparative chemotherapy for the transplant and two days after the last dose of chemotherapy, participants will have allogenic HSCT using the donated stem cells.
* Participants will receive an infusion of NK cells on days 7 and 35 after the HSCT. - Participants will remain in the hospital for monitoring after the HSCT and NK cell treatments, and will be followed closely as outpatients for the first 6 months after the transplant and then less frequently for at least 5 years.

DETAILED DESCRIPTION:
Background

* Despite progress in pediatric oncology, some patient subsets with hematologic malignancies and pediatric solid tumors continue to experience extremely poor overall survival. Allogeneic Hematopoietic Stem Cell Transplant (HSCT) is effective in some high-risk hematologic malignancies.
* Allogeneic HSCT can be performed safely in these patient populations, but disease recurrence is common and new approaches to enhance the antitumor effect of this therapy are needed. Natural killer (NK) mediated killing appears to confer improved outcomes after HSCT for patients with acute myelogenous leukemia (AML) and acute lymphoblastic leukemia (ALL), and NK cell infusions have induced complete remissions in patients with AML.
* Preclinical data demonstrates that activated NK cells readily kill pediatric solid tumors and leukemias, that large numbers of activated NK cells can be generated ex vivo using artificial antigen-presenting cells (APCs) and that the post-transplant period may be favorable for expansion and survival of adoptively transferred NK cells.

Objectives

* To assess the feasibility and toxicity of infusing escalating doses of donor-derived activated NK cell donor lymphocyte infusions (NK-DLI) on Days 7 plus or minus 2 days and 49 plus or minus 7 days following human leukocyte antigen (HLA)-matched T cell depleted (TCD) peripheral blood stem cell transplant (PBSCT) in patients with metastatic or recurrent pediatric solid tumors and high risk leukemias who have unrelated donors or related donors;
* To determine if patients treated in this manner experience rapid, sustained donor engraftment and acceptable rates of acute graft versus host disease (aGVHD) (less than 25% incidence of grade III or grade IV).

Eligibility

-Patients 4-35 years with hematologic malignancies (e.g., ALL, AML, Chronic Myelogenous Leukemia (CML), Hodgkins Lymphoma (HD), Non-Hodgkins Lymphoma (NHL), with a 5/6 or 6/6 HLA-matched related or 9/10 or 10/10 HLA matched unrelated donor.

Design

* Pre-transplant disease specific immune depleting chemotherapy and the preparative regimen will be the same as that used previously on 02-C-0259 and 01-C-0125, for those patients undergoing reduced intensity transplant.
* For patients with ALL or AML, a myeloablative regimen based on current Children's Oncology Group (COG) standard-of- care preparative regimen will also be included.
* Donors will undergo 1-3 apheresis sessions for filgrastim mobilized peripheral blood stem cells (PBSC). This product will be T cell and NK cell depleted prior to cryopreservation. NK cells selected from the product will be used for ex vivo activation and expansion using KT64.4-BBL artificial antigen presenting cells.
* A phase 1 cell dose escalation of donor derived NK-DLI will be performed using 3 dose levels (1 x 10(5), 1 x 10(6) and 1 x 10(7) NK cells/kg) infused on days 21 more or less 3 post-PBSCT and a second infusion on day 49 more or less 7 post-PBSCT.
* Three patients will be enrolled at each dose level, with the cohort expanded to 6 if dose-limiting toxicity occurs. An expanded group of 12 patients will be treated at the highest dose level tolerated.

ELIGIBILITY:
* INCLUSION CRITERIA: PATIENTS (RECIPIENT)
* Hematologic Malignancies Diagnoses:

  1. Acute lymphoblastic leukemia (ALL) with a history of bone marrow relapse in clinical remission (CR) #2 or greater, or in CR#1 if prior induction failure; or with an M1 marrow if unable to achieve CR.
  2. Philadelphia chromosome positive ALL patients who;

     1. Have progressed through or relapsed following tyrosine kinase inhibitor (TKI) therapy or conventional myeloablative therapy

        OR
     2. Are ineligible to receive tyrosine kinase inhibitor (TKI) therapy AND myeloablative hematopoietic stem cell transplant (HSCT)
  3. Acute Myelogenous Leukemia (AML) with a history of bone marrow relapse in remission CR #2 or greater; or with an M1 marrow if unable to achieve CR; or in CR#1 if prior induction failure; or any of the following High-Risk categories:

     1. Fms-related tyrosine kinase 3 (FLT3)/internal tandem duplication (ITD)+ with high allelic ratio > 0.4 (high allelic ration (HR) FLT3/ITD+) regardless of low risk features.
     2. Presence of monosomy 7, monosomy 5, or del5q, without inv(16)/t(16;16) or t(8;21) cytogenetics or NPM or CEBP(alpha) mutations.
     3. Acute myelogenous leukemia (AML) without inv(16)/t(16;16), t(8;21), nucleophosmin (NPM), CCAAT/enhancer binding protein (CEPB)(alpha) mutations, monosomy 7, monosomy 5, del5q, or HR FLT3/ITD+, but with evidence of residual AML (greater than or equal to 0.1%) at end of Induction I.
  4. Hodgkin's and Non-Hodgkin's Lymphoma with refractory disease or relapse after at least one salvage regimen, or after autologous stem cell transplant
  5. Juvenile Myelocytic Leukemia (JMML) with less than 10% blasts in marrow and blood, who are not eligible for effective standard therapies.
* Age: 4 to less than or equal to 35 years old at the time of enrollment for solid tumor patients and 4 to less than or equal to 35 years old for hematologic malignancies.
* All previous cytotoxic chemotherapy must be completed at least 3 weeks prior to study entry. Any prior non-hematologic vital organ toxicity (cardiac, pulmonary, hepatic, renal) of any previous therapy must have resolved to grade 1 or less, unless specified elsewhere in Inclusion Criteria for Patient (Recipient).

EXCEPTIONS:

There is no time restriction in regard to prior intrathecal chemotherapy provided there is complete recovery from any acute toxic effects; or

Subjects receiving standard acute lymphoblastic leukemia (ALL) maintenance chemotherapy will not require washout.

* All previous immunologic or molecularly targeted therapy must be completed at least 1 week prior to study entry. Any prior non-hematologic toxicity of any previous therapy must have resolved to grade 1 or less, unless specified elsewhere in Inclusion Criteria for Patient (Recipient).
* Prior investigational therapy must be completed at least 30 days prior to study entry
* Patients with prior autologous or allogeneic transplant are eligible. Patients must be greater than 100 days post transplant and have no evidence of active graft versus host disease (GVHD).
* Performance status: Eastern Cooperative Oncology Group (ECOG) 0, 1 or 2, or for children less than or equal to 10 years of age, Lansky greater than or equal to 60. Life expectancy greater than 3 months.
* Availability of human leukocyte antigen (HLA)-matched (5-6/6 antigen or 8/8 allele) related or unrelated donor.
* Cardiac function: Left ventricular ejection fraction greater than or equal to 45% by multi-gated acquisition scan (MUGA) or echocardiogram (ECHO), fractional shortening greater than or equal to 28% by ECHO.
* Pulmonary function: Diffusing capacity of the lungs for carbon monoxide (DLCO) >= 40% of the expected value corrected for alveolar volume and hgb for reduced intensity transplant and DLCO >=55% for myeloablative regimen. For children who are unable to cooperate for pulmonary function tests (PFTs), the criterion is: No evidence of dyspnea at rest, no exercise intolerance, and no requirement for supplemental oxygen therapy.
* Liver function: Serum total bilirubin less than 2 mg/dl, serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 2.5 times upper limit of normal. Patients with Gilbert syndrome are excluded from the requirement of a normal bilirubin. (Gilbert syndrome is found in 3-10% of the general population, and is characterized by mild, chronic unconjugated hyperbilirubinemia in the absence of liver disease or overt hemolysis).
* Renal function: Age-adjusted normal serum creatinine according to the following, or a creatinine clearance greater than or equal to 60 ml/min/1.73 m(2):

  * For age (years) of less than or equal to 5, a Maximum serum creatinine (mg/dl) of 0.8
  * For age (years) of greater than 5 but less than or equal to 10, a Maximum serum creatinine (mg/dl) of 1.0
  * For age (years) of greater than 10 but less than or equal to 15, a Maximum serum creatinine (mg/dl) of 1.2
  * For age (years) of greater than 15, a Maximum serum creatinine (mg/dl) of 1.5
* Marrow function: Absolute neutrophil count (ANC) must be greater than 750/mm(3) (unless due to underlying disease in which case there is no grade restriction), platelet count must be greater than or equal to 75,000/mm(3) (not achieved by transfusion) unless due to underlying disease in which case there is no grade restriction). Lymphopenia, cluster of differentiation 4 (CD4) lymphopenia, leukopenia, and anemia will not render patients ineligible.
* Ability to give informed consent. For patients less than 18 years of age their legal guardian must give informed consent. Pediatric patients will be included in age-appropriate discussion in order to obtain verbal assent.

  * Durable power of attorney form completed (patients greater than or equal to 18 years of age only).
  * Female patients (and when relevant their male partners) must be willing to practice birth control (including abstinence) during and for two months after treatment, if of childbearing potential.

EXCLUSION CRITERIA: PATIENT (RECIPIENT)

* Uncontrolled infection.
* Active central nervous system (CNS) malignancy as defined by:

  1. Solid Tumors: History of untreated CNS tumor involvement. Extradural masses which have not invaded the brain parenchyma or parameningeal tumors without evidence for leptomeningeal spread will not render the patient ineligible. Patients with previous CNS tumor involvement are eligible IF the CNS tumor(s) has been treated and has been stable or resolving for at least 6 months; and if the patient does not currently require steroids.
  2. Lymphoma: tumor mass on computed tomography (CT) scan or leptomeningeal disease
  3. Leukemia: CNS 2 or CNS 3 classification.
* Lactating or pregnant females (due to risk to fetus or newborn).
* Human immunodeficiency virus (HIV) positive (due to unacceptable risk associated with severe immune suppression).
* Hepatitis B surface antigen (HBsAg) positive or hepatitis C antibody positive with elevated liver transaminases. All patients with chronic active hepatitis (including those on treatment) are ineligible.
* Patients who require systemic corticosteroid or other immunosuppressive therapy. Immunosuppressive therapy must be stopped at least 28 days prior to protocol cycle 1, day 1 (C1D1). Topical agents and/or inhaled corticosteroids are permitted.
* High risk of inability to comply with transplant protocol, or inability to give appropriate informed consent in the estimation of the principal investigator (PI), social work, psychiatry, or the stem cell transplant team.
* Fanconi Anemia
* Clinically significant systemic illness (e.g. serious active infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), that in the judgment of the PI would likely compromise the patients ability to tolerate protocol therapy or significantly increase the risk of complications.

INCLUSION CRITERIA: DONOR

* Weight greater than or equal to 15 kilograms and for unrelated donors, greater than or equal to 18 years.
* HLA-matched related or unrelated allogeneic donors. Genotypically identical twins may serve as stem cell donors. Related donors must be 5 or 6/6 antigen matched. Unrelated donors must be 8/8 allele matched.
* For donors less than 18 years of age, he/she must be the oldest suitable donor, their legal guardian must give informed consent, the donor must give verbal assent, and he/she must be cleared by social work and a mental health specialist to participate.
* For donors greater than or equal to 18 years of age, ability to give informed consent.
* Adequate peripheral venous access for apheresis or consent to use a temporary central venous catheter for apheresis.
* Donor selection will be in accordance with National Institutes of Health (NIH)/Clinical Center (CC) Department of Transfusion Medicine (DTM) criteria and, in the case of an unrelated donor, the National Marrow Donor Program (NMDP) standards and Food and Drug Administration (FDA) 21 Code of Federal Regulations (CFR) 1271.

EXCLUSION CRITERIA: DONOR

* History of medical illness that in the estimation of the PI or DTM/NMDP physician poses prohibitive risk to donation including, but not limited to, stroke, hypertension that is not controlled with medication, or heart disease. Individuals with symptomatic angina or a history of coronary bypass grafting or angioplasty will not be eligible.
* Anemia (Hemoglobin (Hb) less than 11 gm/dl) or thrombocytopenia (less than100,000/microliters).
* Identical twins will be excluded; the lack of Major histocompatibility complex Major histocompatibility complex (MHC) incompatibility will alter the toxicity profile in such a way as to make the results uninterpretable.
* Breast feeding or pregnant females. Donors of childbearing potential must use an effective method of contraception during the time they are receiving filgrastim. The effects of cytokine administration on a fetus are unknown and may be potentially harmful. The effects upon breast milk are also unknown and may potentially be harmful to the infant.
* High risk of inability to comply with protocol requirements as determined by the principal investigator and donor center team.
* Positive screening test for transfusion-transmissible infection in accordance with DTM or NMDP donation standards, including HIV-positive, hepatitis B surface antigen (HBsAg) positive or hepatitis C antibody positive.

Ages: 4 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2011-01-29 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nirali N Shah, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shah NN, Baird K, Delbrook CP, Fleisher TA, Kohler ME, Rampertaap S, Lemberg K, Hurley CK, Kleiner DE, Merchant MS, Pittaluga S, Sabatino M, Stroncek DF, Wayne AS, Zhang H, Fry TJ, Mackall CL. Acute GVHD in patients receiving IL-15/4-1BBL activated NK cells following T-cell-depleted stem cell transplantation. Blood. 2015 Jan 29;125(5):784-92. doi: 10.1182/blood-2014-07-592881. Epub 2014 Dec 1. PMID 25452614
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0073.html

RESULTS

PARTICIPANT FLOW:
Groups:
- SG1 - Patients With Related Donors at DL1 (1x10^5 Cells/kg): All patients with related donors who received Pre-bone marrow transplant (BMT) Prep Regimen with Peripheral Blood Stem Cell infusion and at least one Natural Killer (NK) cell infusion at a dose of 1x10^5 NK cells/kg.
- SG2 - Patients With Related Donors at DL2 (1x10^6 Cells/kg): All patients with related donors who received Pre-bone marrow transplant (BMT) Prep Regimen with Peripheral Blood Stem Cell infusion and at least one Natural Killer (NK) cell infusion at a dose of 1x10^6 NK cells/kg.
- SG3 - Patients With Unrelated Donors at DL1 (1x10^5 Cells/kg): All patients with unrelated donors who received Pre-bone marrow transplant (BMT) Prep Regimen with Peripheral Blood Stem Cell infusion and at least one Natural Killer (NK) cell infusion at a dose of 1x10^5 NK cells/kg.
- SG4 - Related Donors: All related stem cell donors who received at least one dose of filgrastim for NK cell mobilization.
Period: Overall Study
Arm/Group | SG1 - Patients With Related Donors at DL1 (1x10^5 Cells/kg) | SG2 - Patients With Related Donors at DL2 (1x10^6 Cells/kg) | SG3 - Patients With Unrelated Donors at DL1 (1x10^5 Cells/kg) | SG4 - Related Donors
Started | 4 | 7 | 12 | 11
Completed | 3 | 2 | 5 | 8
Not Completed | 1 | 5 | 7 | 3
Not completed — Patient developed progressive disease | 1 | 1 | 3 | 2
Not completed — Donor anaphylaxis | 0 | 1 | 0 | 1
Not completed — Developed GVHD or complications of BMT | 0 | 1 | 4 | 0
Not completed — Low donor chimerism | 0 | 1 | 0 | 0
Not completed — NK cells did not meet release criteria | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SG1 - Patients With Related Donors at DL1 (1x10^5 Cells/kg) | SG2 - Patients With Related Donors at DL2 (1x10^6 Cells/kg) | SG3 - Patients With Unrelated Donors at DL1 (1x10^5 Cells/kg) | SG4 - Related Donors | Total
Number analyzed (Participants) | 4 | 7 | 12 | 11 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 3 | 5 | 3 | 13
  Between 18 and 65 years | 2 | 4 | 7 | 8 | 21
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 21.4 [14.4 to 33.4] | 21.2 [9.2 to 30.5] | 18.8 [6.2 to 34.5] | 18.9 [12.5 to 30.6] | 18.92 [6.2 to 34.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 1 | 7 | 12
  Male | 4 | 3 | 11 | 4 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3 | 3 | 9
  Not Hispanic or Latino | 4 | 4 | 9 | 8 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2 | 4
  White | 3 | 5 | 9 | 8 | 25
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 7 | 12 | 11 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Received 2 Doses of Natural Killer (NK) Cell Infusions
Description: Participants received 2 doses of natural killer infusions within 56 days of hematopoietic stem cell transplant (HSCT).
Time Frame: within 56 days of hematopoietic stem cell transplant (HSCT)
Population: This outcome measure does not apply to donors as they did not receive the treatment intervention. Two participants in SG2 and three participants in SG3 were not analyzed because they did not receive a transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | SG1 - Patients With Related Donors at DL1 (1x10^5 Cells/kg) | SG2 - Patients With Related Donors at DL2 (1x10^6 Cells/kg) | SG3 - Patients With Unrelated Donors at DL1 (1x10^5 Cells/kg)
Number analyzed (Participants) | 4 | 5 | 9
Participants | 3 | 2 | 5

2. Primary Outcome: Number of Patients Who Received the Highest Dose Level of NK Cells (1x10^6 NK Cells/kg for Patients With Related Donors and 1 x10^5 NK Cells/kg for Patients With Unrelated Donors) With Sustained Donor Lymphoid Engraftment
Description: Donor engraftment is defined as >95% donor lymphoid chimerism (cluster of differentiation 3+T-cells on peripheral blood).
Time Frame: 100 days
Population: This outcome measure does not apply to donors as they did not receive the treatment intervention. Three patients in SG2 where not included because they did not receive any NK cell infusions. Four patients in SG3 were not included because they did not receive any NK cell infusions.
Measure: Count of Participants; unit: Participants
Groups:
- SG3 - Patients With Unrelated Donors at Dose Level 1 (1x10^5 c: All patients with unrelated donors who received Pre-bone marrow transplant (BMT) Prep Regimen with Peripheral Blood Stem Cell infusion and at least one Natural Killer (NK) cell infusion at a dose of 1x10^5 NK cells/kg.
Arm/Group | SG2 - Patients With Related Donors at DL2 (1x10^6 Cells/kg) | SG3 - Patients With Unrelated Donors at Dose Level 1 (1x10^5 c
Number analyzed (Participants) | 4 | 8
Participants | 1 | 5

3. Secondary Outcome: Number of Participants With Mild, Moderate and/or Severe Chronic Graft Versus Host Disease (cGVHD)
Description: Chronic graft versus host disease was assessed by the National Institutes of Health Consensus Criteria. Severity is rated mild moderate or severe on a scale of 0 (no symptoms) -3 (severe symptoms) . Mild is signs and symptoms that do not interfere substantially with function and do not progress once appropriately treated with local therapy. Moderate is signs and symptoms interfere somewhat with function despite appropriate therapy. Severe is signs and symptoms limit function substantially despite appropriate therapy. Low grade is best outcome and high grade is worse outcome.
Time Frame: up to 3 years post-transplant
Population: This outcome measure does not apply to donors as they did not receive the treatment intervention. Three participants in SG2 and four participants in SG3 were not analyzed because they did not receive any NK cell infusions.
Measure: Count of Participants; unit: Participants
Arm/Group | SG1 - Patients With Related Donors at DL1 (1x10^5 Cells/kg) | SG2 - Patients With Related Donors at DL2 (1x10^6 Cells/kg) | SG3 - Patients With Unrelated Donors at DL1 (1x10^5 Cells/kg)
Number analyzed (Participants) | 4 | 4 | 8
Participants
  Mild | 0 | 0 | 2
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

4. Secondary Outcome: Disease-free Survival
Description: Disease free survival is defined as the time interval from start of treatment to documented evidence of disease progression. Progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Progressive disease is at least a 20% increase in the sum of the longest diameter of all target lesions.
Time Frame: 12 months post-transplant
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- SG1 - Patients With Related Donors: All patients with related donors who received Pre-bone marrow transplant (BMT) Prep Regimen with Peripheral Blood Stem Cell infusion and at least one Natural Killer (NK) cell infusion at a dose of 1x10^5 NK cells/kg.
- SG2 - Patients With Unrelated Donors: All patients with related donors who received Pre-bone marrow transplant (BMT) Prep Regimen with Peripheral Blood Stem Cell infusion and at least one Natural Killer (NK) cell infusion at a dose of 1x10^6 NK cells/kg.
Arm/Group | SG1 - Patients With Related Donors | SG2 - Patients With Unrelated Donors | SG3 - Patients With Unrelated Donors at DL1 (1x10^5 Cells/kg)
Number analyzed (Participants) | 4 | 4 | 8
Months | 2.8 [1.8 to 3.1] | 8.7 [2 to 12] | 10.35 [6.2 to 12]

5. Secondary Outcome: Overall Survival Since Date of Transplant
Description: Overall survival is defined as the time from date of transplant until date of death or date last known alive.
Time Frame: Up to 36 months post-transplant
Population: This outcome measure does not apply to donors as they did not undergo transplant. Three participants in SG2 and four participants in SG3 were not analyzed because they did not receive any NK cell infusions.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | SG1 - Patients With Related Donors at DL1 (1x10^5 Cells/kg) | SG2 - Patients With Related Donors at DL2 (1x10^6 Cells/kg) | SG3 - Patients With Unrelated Donors at DL1 (1x10^5 Cells/kg)
Number analyzed (Participants) | 4 | 4 | 8
Months | 15.5 [5.8 to 30.2] | 34 [6.3 to 36] | 10.5 [6.4 to 36]

6. Secondary Outcome: Number of Occurrences of Viral Infection and/or Reactivation in Allogeneic Peripheral Blood Stem Cell Transplant (PBSCT) Followed by Natural Killer-donor Lymphocyte Infusion (NK-DLI)
Description: One or more occurrences of a new infection, reactivation or both (e.g. cytomegalovirus + flu, for example). Viral infections increase a patient's risk for a worse outcome and viral reactivation is a marker for T-cell immune dysregulation (i.e., inflammation).
Time Frame: Within 1-year post-transplant
Population: as for outcome 3
Measure: Number; unit: viral infections/reactivations
Groups:
- SG2 - Patients With Related Donors at DL 2 (1x10^6 Cells/kg): All patients with related donors who received Pre-bone marrow transplant (BMT) Prep Regimen with Peripheral Blood Stem Cell infusion and at least one Natural Killer (NK) cell infusion at a dose of 1x10^6 NK cells/kg.
Arm/Group | SG1 - Patients With Related Donors at DL1 (1x10^5 Cells/kg) | SG2 - Patients With Related Donors at DL 2 (1x10^6 Cells/kg) | SG3 - Patients With Unrelated Donors at Dose Level 1 (1x10^5 c
Number analyzed (Participants) | 4 | 4 | 8
viral infections/reactivations | 6 | 11 | 14

7. Secondary Outcome: Number of Participants With a Decline in Interleukin 7 (IL-7) and Interleukin 15 (IL-15) Cell Numbers Post-Transplant
Description: Cytokine levels are checked in a multiplex format according to manufacturer's instructions (Meso Scale Discovery, Gaithersburg, Maryland, United States of America (USA).
Time Frame: 3 years
Population: This outcome measure was not performed.The data was not collected for this outcome measure because the original Principal Investigator departed the institution. The protocol was transferred to a new Principal Investigator who elected not to pursue this outcome.
Arm/Group | SG1 - Patients With Related Donors at DL1 (1x10^5 Cells/kg) | SG2 - Patients With Related Donors at DL2 (1x10^6 Cells/kg) | SG3 - Patients With Unrelated Donors at DL1 (1x10^5 Cells/kg)
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Presence of Killer-cell Immunoglobulin-like Receptors (KIR) Gene Mismatch
Description: Blood samples and/or buccal swabs were obtained and the presence of Killer-cell immunoglobulin-like receptors (KIR) genes was determined by locus specific polymerase chain reaction (PCR) amplification followed by gel electrophoresis. KIR receptors were examined for a mismatch in the human leukocyte antigen (HLA) ligand. A mismatch in the HLA ligand can signal increased anti-tumor activity, enhanced engraftment, and/or less infectious complications for patients.
Time Frame: Prior to stem cell transplant (Day 0)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | SG1 - Patients With Related Donors at DL1 (1x10^5 Cells/kg) | SG2 - Patients With Related Donors at DL 2 (1x10^6 Cells/kg) | SG3 - Patients With Unrelated Donors at DL1 (1x10^5 Cells/kg)
Number analyzed (Participants) | 4 | 4 | 8
Participants | 3 | 2 | 5

9. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned
Time Frame: Date treatment consent signed to date off study, approximately 65 months and 2 days.
Measure: Count of Participants; unit: Participants
Arm/Group | SG1 - Patients With Related Donors at DL1 (1x10^5 Cells/kg) | SG2 - Patients With Related Donors at DL2 (1x10^6 Cells/kg) | SG3 - Patients With Unrelated Donors at DL1 (1x10^5 Cells/kg) | SG4 - Related Donors
Number analyzed (Participants) | 4 | 7 | 12 | 11
Participants | 4 | 7 | 12 | 8

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 65 months and 2 days.
Description: The majority of participants listed in All-Cause Mortality died from progressive disease. There were two patients who died from transplant-related complications.
Arm/Group | SG1 - Patients With Related Donors at DL1 (1x10^5 Cells/kg) | SG2 - Patients With Related Donors at DL2 (1x10^6 Cells/kg) | SG3 - Patients With Unrelated Donors at DL1 (1x10^5 Cells/kg) | SG4 - Related Donors
All-Cause Mortality (participants affected / at risk) | 4/4 | 6/7 | 8/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/4 | 4/7 | 6/12 | 1/11
Other Adverse Events (participants affected / at risk) | 4/4 | 7/7 | 12/12 | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SG1 - Patients With Related Donors at DL1 (1x10^5 Cells/kg) (N=4) | SG2 - Patients With Related Donors at DL2 (1x10^6 Cells/kg) (N=7) | SG3 - Patients With Unrelated Donors at DL1 (1x10^5 Cells/kg) (N=12) | SG4 - Related Donors (N=11)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylaxis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (6) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Eye disorders - Other, CMV Retinitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
GGT increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hepatic hemorrhage (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hepatic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other, Liver ( GVHD) (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, CMV reactivation (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Infections and infestations - Other, PCP Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Salmonella in stool (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Infections and infestations - Other, c difficile positive (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — - Other, Hilar cholangiocarcinoma
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal hemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SG1 - Patients With Related Donors at DL1 (1x10^5 Cells/kg) (N=4) | SG2 - Patients With Related Donors at DL2 (1x10^6 Cells/kg) (N=7) | SG3 - Patients With Unrelated Donors at DL1 (1x10^5 Cells/kg) (N=12) | SG4 - Related Donors (N=11)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 5 (13) | 6 (13) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (2) | 3 (12) | 9 (16) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Akathisia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (9) | 6 (50) | 11 (64) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 2 (4) | 2 (4) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 3 (3) | 5 (6) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Anal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 4 (31) | 7 (85) | 9 (108) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (4) | 6 (16) | 11 (24) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (6) | 4 (6) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (15) | 5 (47) | 9 (70) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (7) | 6 (18) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, Diffusely edematous (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, varicose veins (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (5) | 3 (19) | 5 (17) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 4 (6) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (7) | 3 (4) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 5 (10) | 3 (4) | 1 (1)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
CPK increased (Investigations) | 1 (3) | 2 (4) | 4 (4) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 2 (2) | 2 (3) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (3) | 1 (2) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Chills (General disorders) | 4 (6) | 3 (5) | 6 (9) | 0 (0)
Cholesterol high (Investigations) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 3 (7) | 4 (8) | 0 (0)
Corneal ulcer (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (6) | 10 (18) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 2 (5) | 6 (26) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 2 (4) | 2 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (7) | 4 (12) | 9 (45) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 3 (6) | 5 (10) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 3 (4) | 8 (9) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (7) | 9 (13) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 5 (7) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Edema face (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 2 (6) | 5 (5) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (6) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Eye disorders - Other, Amblyopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye disorders - Other, double vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye disorders - Other, ocular GVHD (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye disorders - Other, keratopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Eyelid function disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (8) | 5 (9) | 5 (10) | 1 (1)
Fever (General disorders) | 4 (14) | 3 (9) | 11 (88) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (8) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
GGT increased (Investigations) | 0 (0) | 1 (6) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (3) | 3 (3) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
General disorders and administration site conditions - Other, Anasarca (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, edema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, generalized edema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gum infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Haptoglobin decreased (Investigations) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 6 (28) | 8 (28) | 4 (5)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Hematuria (Renal and urinary disorders) | 2 (6) | 1 (3) | 3 (9) | 0 (0)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Venous occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hepatobiliary disorders - Other, intrahepatic biliary ductal stricture (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 3 (9) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (38) | 6 (82) | 12 (160) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 4 (8) | 4 (4) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 2 (6) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (4) | 4 (12) | 6 (22) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (2) | 1 (3) | 5 (7) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 3 (3) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (25) | 5 (33) | 10 (92) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (39) | 5 (26) | 11 (157) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (9) | 0 (0) | 3 (17) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (5) | 6 (15) | 7 (45) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 5 (29) | 8 (112) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 5 (17) | 8 (29) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (18) | 4 (30) | 10 (99) | 0 (0)
Hypotension (Vascular disorders) | 2 (4) | 3 (5) | 5 (14) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Immune system disorders - Other, red man syndrome with vanco (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Adenovirus viremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, C. diff infection (Infections and infestations) | 2 (2) | 2 (3) | 1 (1) | 0 (0)
Infections and infestations - Other, cytomegalovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Infections and infestations - Other, E. coli bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Enterococcus faecalis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, Gram Positive (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, salmonella positive (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, upper respiratory infection (Infections and infestations) | 0 (0) | 3 (3) | 4 (5) | 0 (0)
Infections and infestations - Other, urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 5 (7) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 2 (14) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - Other, bicarbonate, low (Metabolism and nutrition disorders) | 2 (3) | 5 (27) | 8 (54) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (4) | 5 (11) | 8 (18) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, hand stiff (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, wrist weakness bilaterally (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (6) | 3 (8) | 0 (0) | 3 (3)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (15) | 5 (29) | 8 (32) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (5) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (51) | 7 (96) | 12 (107) | 3 (3)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pain (General disorders) | 1 (3) | 5 (24) | 6 (17) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Periorbital edema (Eye disorders) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Peritoneal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 4 (43) | 6 (97) | 12 (239) | 6 (10)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 5 (5) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Proteinuria (Renal and urinary disorders) | 3 (12) | 2 (4) | 5 (45) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 5 (13) | 7 (16) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (4) | 4 (9) | 9 (43) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 5 (6) | 0 (0)
Renal and urinary disorders - Other, bladder spasm intermittent (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, renal proximal tubular damage (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, trouble maintaining urinary stream (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Reproductive system and breast disorders - Other, urethral irritation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — (crackles on bilateral bases)
Retinal vascular disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Salivary duct inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scrotal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scleral disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Serum amylase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 5 (7) | 7 (9) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Skin and subcutaneous tissue disorders - Other, erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, genital lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Erythema surrounding Hickman (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, hyperkeratotic papules (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (4) | 6 (9) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (4) | 0 (0)
Superficial thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, inguinal pain on surgical site (Surgical and medical procedures) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, jaw inflammation (S/P extraction) (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, pain in the biliary drain (Surgical and medical procedures) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, bleeding from ETT (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 2 (2) | 0 (0) | 3 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Urostomy obstruction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (11) | 5 (20) | 9 (28) | 1 (1)
Watering eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight gain (Investigations) | 0 (0) | 1 (3) | 1 (7) | 0 (0)
Weight loss (Investigations) | 0 (0) | 2 (9) | 9 (63) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 4 (65) | 6 (97) | 12 (176) | 3 (3)
Electrocardiogram QT corrected prolonged (Cardiac disorders) | 1 (4) | 1 (3) | 0 (0) | 0 (0)
Otitis externa (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and Infestations - Other, Bacteremia (Infections and infestations) | 0 (0) | 2 (2) | 3 (5) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alkaline aminotransferase (Investigations) | 0 (0) | 4 (11) | 5 (14) | 2 (2)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (5) | 5 (6) | 6 (8) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/04/NCT01287104/Prot_SAP_000.pdf
  • Informed Consent Form: Standard-Addendum (2016-01-08): https://cdn.clinicaltrials.gov/large-docs/04/NCT01287104/ICF_001.pdf
  • Informed Consent Form: Donor (2016-01-08): https://cdn.clinicaltrials.gov/large-docs/04/NCT01287104/ICF_002.pdf
  • Informed Consent Form: Recipient (2016-01-08): https://cdn.clinicaltrials.gov/large-docs/04/NCT01287104/ICF_003.pdf